CLINICAL TRIAL: NCT05388422
Title: Physical Measurement in Patients With Severe Cerebral Palsy Using 3D Scanner and Improvement of Manufacturing Techniques for Hip Dislocation Prevention Assistive Devices
Brief Title: Application of 3D Scanner to Measure Physical Size in Patients With Severe Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-2201-732-001
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Cerebral Palsy, Spastic
Keywords: 3D Scanner; Cerebral palsy; Hip dislocation; Orthotic devices; Protective devices
MeSH Terms: conditions — Cerebral Palsy; Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe cerebral palsy (GMFCS IV and V) (Experimental): This study included patients with severe cerebral palsy (GMFCS IV and V)
  Interventions: Device: Application of 3D scanner to measure physical size in patients with severe cerebral palsy

INTERVENTIONS:
Device: Application of 3D scanner to measure physical size in patients with severe cerebral palsy — Before starting the study, radiologic and clinical evaluation were performed. After measuring the patient's exact physical size by applying a 3D scanner, we manufacture hip brace in preventing progressive hip displacement in patients with severe cerebral palsy. After wearing for a week, follow-up radiologic and clinical evaluation were performed.

SUMMARY:
The aim of this study is to improve the manufacturing techniques of hip brace in preventing progressive hip displacement in patients with severe cerebral palsy, through the measurement of patient's physical size using a 3D scanner.

DETAILED DESCRIPTION:
1. Design : Prospective Study
2. Setting: Hospital rehabilitation department and Home
3. Intervention: Before starting the study, radiologic and clinical evaluation were performed. After measuring the patient's exact physical size by applying a 3D scanner, we manufacture hip brace in preventing progressive hip displacement in patients with severe cerebral palsy. After wearing for a week, follow-up radiologic and clinical evaluation were performed.
4. Main outcome measure 1) Primary outcome: right, left, both hip MI 2) Secondary outcomes: the hip and knee joint range of motion (ROM), pain intensity, satisfaction and discomfort score for the hip brace, quality of life (QOL) of the patients and their caregivers, and the wearability test.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of cerebral palsy
2. age 1-15 years
3. GMFCS Level IV, V
4. quadriplegia, or diplegia for more than 6 months
5. Patients who have written consent with permission from the child and caregiver.

Exclusion Criteria:

1. Patients who did not agree to participate in the study
2. Patients who refused the examination
3. Patients who had hip surgery experience
4. Patients who were scheduled to undergo surgery during the clinical study
5. Patients who could not be measured with a 3D scanner

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Migration index | 1 weeks
  Hip AP radiography

SECONDARY OUTCOMES:
Visual analog scale (Pain index) | 1 weeks
  measure the pain expressed by score from 0 to 10. The closer to 10, the higher the pain.
Caregiver Priorities & Child Health Index of Life with Disabilities (CPCHILD) | 1 weeks
  measure the quality of life expressed by score from 0 to 100. The higher the quality of life.
Likert scale (score) | 1 weeks
  measure the satisfaction, and discomfort about hip protection orthosis expressed by score from 1 to 5. The closer to 1, the higher the satisfaction or comfort.
Range of motion of hip joint | 1 weeks
  Using goniometer, measure the hip and knee abduction and flexion angle expressed by degree from 0' to 180'. The closer to 180', the better the value.
wearability test | 1 weeks
  the Wearability Test consisted of four questions on wearing sensation, five questions about on fit, and four questions on motion suitability evaluation. Each item was scored on 5-point scale, with a total score of 65.

CONTACTS AND LOCATIONS:
Overall Officials: Juseok Ryu, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University Bundang Hospital, Seoul National University College of Medicine, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim JM, Lim J, Choi SY, Rhim SH, Beom J, Ryu JS. Application of 3D scanner to measure physical size and improvement of hip brace manufacturing technology in severe cerebral palsy patients. Sci Rep. 2023 Nov 24;13(1):20691. doi: 10.1038/s41598-023-47665-w. PMID 38001232